CLINICAL TRIAL: NCT02331576
Title: Femoral Nerve Block in Patient With Total Knee Arthroplasty; Analgesic Effect of Perineural Fentanyl Additive to Local Anesthetics
Brief Title: Analgesic Effect of Perineural Fentanyl Additive to Local Anesthetics in Femoral Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, BHeo, assistant professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNUHH-2014-141
Record Dates: First submitted 2014-12-23; First posted 2015-01-06 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rocaine (Placebo Comparator): continuous femoral nerve block with ropivacaine alone.
  Interventions: Drug: rocaine
- rocaine with fentanyl (Active Comparator): continuous femoral nerve block with combination of ropivacaine and fentanyl.
  Interventions: Drug: rocaine; Drug: Fentanyl

INTERVENTIONS:
Drug: rocaine
  Other Names: ropivacaine HCL
Drug: Fentanyl
  Other Names: fentanyl citrate
  Arms: rocaine with fentanyl

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy of perineural fentanyl combined with local anesthetics in the post operative pain control with continuous femoral nerve block after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients who scheduled to receive knee arthroplasty with general anesthesia
* ASA physical status 1 or 2

Exclusion Criteria:

* allergy to drug
* refuse to the study
* ASA physical status 3 and 4
* history of drug abuse
* cognitive disfunction such as dementia
* patients who do not adequate for general anesthesia

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogue Scales by time sequence | baseline(just after operation), 15, 30, 60 minute and 24 hour after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bongha Heo, Dr, Principal Investigator — assistant professor
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea